CLINICAL TRIAL: NCT01081717
Title: A Large US Health Insurance Claims Database Will be Used to Estimate the Incidence of Serious Outcomes in Patients With Rheumatoid Arthritis, Psoriatic Arthritis, or Ankylosing Spondylitis Treated With Golimumab and Other Types of Biological and Systemic Non Biological Treatments
Brief Title: Golimumab Safety and Surveillance Program Using the Ingenix NHI Database
Status: Completed | Type: Observational
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016720; CNTO148ART4002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis; Arthritis, Psoriatic; Ankylosing Spondylitis
Keywords: Rheumatoid arthritis; psoriatic arthritis; ankylosing spondylitis; golimumab; anti-TNF biologics; non-anti-TNF biologics; non-biological treatments
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing | interventions — golimumab; Sociology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 001: golimumab as prescribed
  Interventions: Biological: golimumab
- 002: anti-TNF biologics as prescribed
  Interventions: Biological: anti-TNF biologics
- 003: non-anti-TNF biologics as prescribed
  Interventions: Biological: non-anti-TNF biologics
- 004: systemic non-biological treatments as prescribed
  Interventions: Drug: systemic non-biological treatments
- 005: general population non-treated cohort
  Interventions: Other: general population

INTERVENTIONS:
Drug: systemic non-biological treatments — as prescribed
  Groups: 004
Biological: anti-TNF biologics — as prescribed
  Groups: 002
Biological: golimumab — as prescribed
  Groups: 001
Biological: non-anti-TNF biologics — as prescribed
  Groups: 003
Other: general population — non-treated cohort
  Groups: 005

SUMMARY:
The participants included in this observational study will be drawn from a research database containing claims and enrollment data for members of a large, geographically diverse US health plan.The objective of this study is to estimate the rate of serious infections, tuberculosis, malignancies, and other outcomes in rheumatoid arthritis, psoriatic arthritis, and ankylosing spondylitis patients treated with golimumab, anti-tumor necrosis factor (TNF) biologics, non-anti-TNF biologics, or systemic non-biological treatments.

DETAILED DESCRIPTION:
The participants included in this study will be drawn from the Ingenix Normative Health Informatics Database, a proprietary research database containing claims and enrollment data dating back to 1993 for members of a large, geographically diverse US health plan. This study will include cohorts of participants who have claims consistent with a diagnosis of rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis and who initiate golimumab, anti-TNF biologics, non-anti-TNF biologics, or systemic non-biological treatments. Participants will be identified by claims bearing codes for dispensed drugs, procedures or diagnoses and followed after the launch of golimumab for up to 8 years. A sample of enrolled health plan members without claims evidence of diagnosis or treatment of Rheumatoid arthritis, psoriatic arthritis or ankylosing spondylitis will also be selected. The claims database will be used to estimate the incidence of the primary outcomes of serious infections, tuberculosis (TB) and non-TB mycobacterial infections, malignancies such as lymphoma, and other selected outcomes. No study agents will be administered in this study. All participants will receive standard-of-care treatment as prescribed by their physician

ELIGIBILITY:
Inclusion Criteria:

* Complete medical coverage and pharmacy benefits
* Six months of continuous enrollment prior to the date of cohort entry

Exclusion Criteria:

* Participants will be excluded if they do not have information on age, gender or enrollment

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include cohorts of patients who have claims consistent with a diagnosis of rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis who initiate golimumab, anti-TNF biologics, non-anti-TNF biologics, or systemic non-biological treatments, within the Ingenix Normative Health Informatics Database.
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2009-04-14 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Estimate incidence of serious infections, malignancies, and other selected outcomes in patients with rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis initiating golimumab and other biological and systemic non-biological treatment | The study will be approximately 8 years in duration

CONTACTS AND LOCATIONS:
Overall Officials: Anja Geldhof, Eng, Ph.D., Study Director — Janssen Biotech, Inc.